CLINICAL TRIAL: NCT05184400
Title: Identification of New Biomarkers for Patients With Biliary Tract Cancer (Cholangiocarcinoma and Gallbladder Cancer) - do They Provide New Information Regarding Diagnosis, Treatment Efficacy, Side Effects, or Prognosis?
Brief Title: Identification of New Biomarkers for Patients With Cholangiocarcinoma and Gallbladder Cancer
Acronym: CHOCA
Status: Recruiting | Type: Observational
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Troels Dreier Christensen, Principal Investigator, Herlev and Gentofte Hospital
Other Study IDs: GI1412
Record Dates: First submitted 2021-10-21; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Biliary Tract Cancer; Cholangiocarcinoma; Gallbladder Cancer
Keywords: Prospective observational open cohort study; Biomarkers; Diagnostics; Prognostics; Prediction of treatment efficacy
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma; Gallbladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (i.e. serum, EDTA plasma and buffy coat, and blood in PAXgeneRNA tubes) are collected from all patients before operation or start of chemotherapy and during treatment with blood sampling before the 2nd cycle of chemotherapy and longitudinally every time of CT scan until disease progression. Tissue removed during routine diagnostic procedures or treatment will be requisitioned.
Oversight: Data Monitoring Committee: No

SUMMARY:
No validated biomarkers exist that can identify patients with biliary tract cancer at an early stage or predict treatment outcomes. The objective of the present study is to find diagnostic, prognostic and predictive biomarkers.

DETAILED DESCRIPTION:
Biliary tract cancer (BTC) is a heterogeneous disease and includes both gallbladder cancer and cholangiocarcinoma. Combined BTC is the fifth most common gastrointestinal cancer. The prognosis is poor with a median overall survival of less than a year and estimated 5-year survival of about 20 % for all stages. The poor survival is related to aggressive malign nature, late diagnosis, and limited treatment options. Today, only CA 19-9 is used in routine practice but its use as a prognostic or diagnostic biomarker is very limited.

The objective of the present study is to find diagnostic, prognostic, and predictive biomarkers, which can be used to 1) diagnose BTC early in the disease course with high specificity and sensitivity, 2) improve prognostication, or 3) predict and monitor treatment effectiveness and tolerability for the individual patient.

CHOCA is an observational and translational open cohort study with a prospective collection of biological materials (blood samples and tissue) and clinical data in patients with BTC receiving standard or protocolized treatment. Blood samples (i.e. serum, EDTA plasma and buffy coat, and blood in PAXgeneRNA tubes) are collected from all patients before operation or start of chemotherapy and during treatment with blood sampling before the 2nd cycle of chemotherapy and longitudinally at the time of follow-up CT scan (about every 3 months) until disease progression. Tissue removed during routine diagnostic procedures or treatment will be requisitioned.

The patients are followed until death. The following data are collected: Demographics, disease characteristics, comorbidities and lifestyle factors, routine blood tests (i.e. hematology, creatinine, liver enzymes, bilirubin, carbohydrate antigen 19-9, C-reactive protein); type of operation; types of chemotherapy, reason for termination of therapy; date of disease recurrence in operated patients; date of disease progression for each line of chemotherapy; and date of death. Biomarker analyses will include a range of molecules with different characteristics such as DNA, Single Nucleotide Polymorphism (SNPs), RNA, microRNA, proteins, proteoglycans, and metabolites. Controls will be included from other studies in order to identify potential diagnostic biomarkers,. Controls include patients with other diseases or healthy subjects. Biomarkers will be analyzed using appropriate methods and statistical analysis following REMARK guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of BTC
* Patients referred for treatment of BTC
* Signed informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients with BTC referred for oncological treatment (adjuvant, neoadjuvant, or palliative setting [any treatment line]) at the Department of Oncology, Herlev & Gentofte Hospital, Denmark and patients referred for surgery at Rigshospitalet (Denmark). The two sites are responsible for all treatment of BTC in eastern Denmark, a region with a population of almost 2.7 million.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy (sensitivity and specificity) | Baseline
  Outcome for diagnostic biomarkers. Case-control design.
Overall survival (OS) | Baseline to death or lost to follow-up, an average of 1 year
  Outcome for prognostic and predictive biomarkers

SECONDARY OUTCOMES:
Progression free survival (PFS) | Baseline to progression, death or lost to follow-up, an average of 1 year
  Outcome for prognostic and predictive biomarkers
Incidence of adverse events | Baseline to progression, death or lost to follow-up, an average of 1 year
  Outcome for prognostic and predictive biomarkers related to treatment toxicity.

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev & Gentofte Hospital, Herlev, Copenhagen, Denmark